CLINICAL TRIAL: NCT02487303
Title: Intravenous Versus Oral Acetaminophen for Postoperative Pain Control After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00041193
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
Keywords: Acetaminophen; Pain, Postoperative; Analgesia, Obstetrical; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetaminophen Intravenous (Active Comparator): (group 1) 1 gram IV acetaminophen every 8 hours for three doses
  Interventions: Drug: Acetaminophen Intravenous
- Acetaminophen Oral (Active Comparator): (group 2) 1 gram oral acetaminophen every 8 hours for three doses
  Interventions: Drug: Acetaminophen Oral
- No acetaminophen (No Intervention): (group 3) no acetaminophen

INTERVENTIONS:
Drug: Acetaminophen Intravenous — IV 1 gram f3 doses over 24 hours
  Other Names: Tylenol
  Arms: Acetaminophen Intravenous
Drug: Acetaminophen Oral — Oral 1 gram 3 doses over 24 hours
  Other Names: Tylenol
  Arms: Acetaminophen Oral

SUMMARY:
This study will compare IV (intravenous) versus oral (PO) acetaminophen for postoperative pain after scheduled, elective Cesarean delivery. All patients will receive a standardized spinal anesthetic for operative anesthesia and will be randomized into one of three groups: (group 1) 1 gram IV acetaminophen every 8 hours for three doses, (group 2) 1 gram oral acetaminophen every 8 hours for three doses, or (group 3) no acetaminophen. This will be a randomized, open label study.

DETAILED DESCRIPTION:
This study will compare IV versus PO acetaminophen for postoperative pain in parturients after scheduled, elective Cesarean delivery. It is designed as a randomized, open label, controlled trial. All patients will receive a standardized spinal anesthetic for operative anesthesia and will be randomized into one of three groups: (group 1) 1 gram IV acetaminophen every 8 hours for three by a computer generated list.

ELIGIBILITY:
Inclusion Criteria:

* Parturients 18 years
* Elective Cesarean delivery
* Spinal anesthesia
* Able to consent to the study and participate in the follow-up.

Exclusion Criteria:

* Weight under 50 kgs
* Allergy to acetaminophen
* General anesthesia
* Urgent or emergent cases
* Bleeding diathesis or other coagulopathy
* G6PD deficiency
* Liver disease
* Substance abuse or dependence
* HELLP syndrome
* Thrombocytopenia or platelet dysfunction
* History or active gastrointestinal bleeding
* Acute kidney injury or chronic renal insufficiency
* Contraindication/refusal to spinal anesthesia
* Chronic pain
* Chronic narcotic use
* Illicit drug use
* Allergy to any study related medications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Result] Macario A, Royal MA. A literature review of randomized clinical trials of intravenous acetaminophen (paracetamol) for acute postoperative pain. Pain Pract. 2011 May-Jun;11(3):290-6. doi: 10.1111/j.1533-2500.2010.00426.x. Epub 2010 Nov 28. PMID 21114616
- [Result] Smith HS. Perioperative intravenous acetaminophen and NSAIDs. Pain Med. 2011 Jun;12(6):961-81. doi: 10.1111/j.1526-4637.2011.01141.x. Epub 2011 May 31. PMID 21627768
- [Result] Wininger SJ, Miller H, Minkowitz HS, Royal MA, Ang RY, Breitmeyer JB, Singla NK. A randomized, double-blind, placebo-controlled, multicenter, repeat-dose study of two intravenous acetaminophen dosing regimens for the treatment of pain after abdominal laparoscopic surgery. Clin Ther. 2010 Dec;32(14):2348-69. doi: 10.1016/j.clinthera.2010.12.011. PMID 21353105
- [Result] Singla NK, Parulan C, Samson R, Hutchinson J, Bushnell R, Beja EG, Ang R, Royal MA. Plasma and cerebrospinal fluid pharmacokinetic parameters after single-dose administration of intravenous, oral, or rectal acetaminophen. Pain Pract. 2012 Sep;12(7):523-32. doi: 10.1111/j.1533-2500.2012.00556.x. Epub 2012 Apr 24. PMID 22524979
- [Result] Fenlon S, Collyer J, Giles J, Bidd H, Lees M, Nicholson J, Dulai R, Hankins M, Edelman N. Oral vs intravenous paracetamol for lower third molar extractions under general anaesthesia: is oral administration inferior? Br J Anaesth. 2013 Mar;110(3):432-7. doi: 10.1093/bja/aes387. Epub 2012 Dec 6. PMID 23220855
- [Result] Alhashemi JA, Alotaibi QA, Mashaat MS, Kaid TM, Mujallid RH, Kaki AM. Intravenous acetaminophen vs oral ibuprofen in combination with morphine PCIA after Cesarean delivery. Can J Anaesth. 2006 Dec;53(12):1200-6. doi: 10.1007/BF03021581. PMID 17142654
- [Result] Wong JY, Carvalho B, Riley ET. Intrathecal morphine 100 and 200 mug for post-cesarean delivery analgesia: a trade-off between analgesic efficacy and side effects. Int J Obstet Anesth. 2013 Jan;22(1):36-41. doi: 10.1016/j.ijoa.2012.09.006. Epub 2012 Nov 15. PMID 23159009
- [Result] Singh SI, Rehou S, Marmai KL, Jones APM. The efficacy of 2 doses of epidural morphine for postcesarean delivery analgesia: a randomized noninferiority trial. Anesth Analg. 2013 Sep;117(3):677-685. doi: 10.1213/ANE.0b013e31829cfd21. Epub 2013 Aug 6. PMID 23921652
- [Result] Beatty NC, Arendt KW, Niesen AD, Wittwer ED, Jacob AK. Analgesia after Cesarean delivery: a retrospective comparison of intrathecal hydromorphone and morphine. J Clin Anesth. 2013 Aug;25(5):379-383. doi: 10.1016/j.jclinane.2013.01.014. Epub 2013 Aug 17. PMID 23965210
- [Derived] Wilson SH, Wolf BJ, Robinson SM, Nelson C, Hebbar L. Intravenous vs Oral Acetaminophen for Analgesia After Cesarean Delivery: A Randomized Trial. Pain Med. 2019 Aug 1;20(8):1584-1591. doi: 10.1093/pm/pny253. PMID 30561704

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
Started | 49 | 51 | 48
Completed | 47 | 47 | 47
Not Completed | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen | Total
Number analyzed (Participants) | 47 | 47 | 47 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 47 | 47 | 141
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.7 [19 to 44] | 30.5 [21 to 43] | 31.2 [18 to 49] | 30.1 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 47 | 141
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 22 | 14 | 21 | 57
  White | 24 | 32 | 26 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 47 | 141

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Postoperative Opiate Consumption
Description: Cumulative opiate consumption (IV morphine equivalents)
Time Frame: 24 hours
Measure: Mean (Full Range); unit: mg
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
Number analyzed (Participants) | 47 | 47 | 47
mg | 2.9 [0 to 28] | 3.8 [0 to 17.5] | 5.7 [0 to 33]

2. Secondary Outcome: Time to First Opiate Rescue
Description: Time to first opiate pain medicine requested by patient
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: hours
Groups:
- Acetaminophen Intravenous: 1 gram IV acetaminophen every 8 hours for three doses
- Acetaminophen Oral: 1 gram oral acetaminophen every 8 hours for three doses
- No Acetaminophen: No acetaminophen
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
Number analyzed (Participants) | 47 | 47 | 47
hours | 25.3 (8.5) | 24.0 (26.3) | 21.3 (23.9)

3. Secondary Outcome: VAS (Visual Analog Scale)
Description: Visual Analog Scale (VAS) pain assessment with ambulation. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]) .
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
Number analyzed (Participants) | 47 | 47 | 47
units on a scale | 37.8 (3.23) | 44.3 (3.28) | 50.8 (3.31)

4. Secondary Outcome: Time Discharge
Description: Time patient meets discharge criteria will be recorded
Time Frame: 24 hours postoperative
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
Number analyzed (Participants) | 47 | 47 | 47
hours | 48.4 (13.7) | 48.6 (11.3) | 50.5 (15.7)

ADVERSE EVENTS:
Time Frame: The timeframe for adverse event data was collected up to 48 hours.
Arm/Group | Acetaminophen Intravenous | Acetaminophen Oral | No Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT02487303/Prot_SAP_000.pdf